CLINICAL TRIAL: NCT01140945
Title: Periodontal Status of Males Attending in Vitro Fertilization Clinic
Brief Title: Association Study Between Periodontal Disease and Male Infertility
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Avigdor Klinger DMD, PhD, Department of Periodontology, Hadassah Medical Organization
Other Study IDs: Klinger-HMO-CTIL
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-01

CONDITIONS: Periodontitis; Sub-fertility
MeSH Terms: conditions — Periodontitis; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Males attending in vitro fertilization clinic

SUMMARY:
The aim of the present study is to examine the association between fertility parameters and the periodontal status of men attending fertility and in vitro fertilization clinic.

DETAILED DESCRIPTION:
An association has been found between periodontal diseases and preterm low birth weight, coronary heart disease, and cerebral infarction. Anaerobic gram negative bacterial plaque that forms subgingivally is the direct causative factor for the development of Gingivitis and Periodontitis.

However, its possible association with male infertility have not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in study

Exclusion Criteria:

* Systemic uncontrolled disease

Ages: 20 Years to 50 Years | Sex: Male
Age Groups: Adult
Study Population: Males attending in vitro fertiliztion clinic
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Positive association between periodontitis and infertility

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical organization, Jerusalem, Israel

REFERENCES:
- [Derived] Klinger A, Hain B, Yaffe H, Schonberger O. Periodontal status of males attending an in vitro fertilization clinic. J Clin Periodontol. 2011 Jun;38(6):542-6. doi: 10.1111/j.1600-051X.2011.01720.x. Epub 2011 Mar 28. PMID 21443558